CLINICAL TRIAL: NCT03375983
Title: Clinical Study of Plasmodium Immunotherapy for Advanced Cancers
Brief Title: Plasmodium Immunotherapy for Advanced Cancers
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CAS Lamvac Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZKLH-003
Record Dates: First submitted 2017-12-10; First posted 2017-12-18 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Advanced Cancers
Keywords: Advanced cancer; Plasmodium immunotherapy; Plasmodiun vivax

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blood-stage infection of P.vivax (Experimental): This is a single arm study that plans to enroll 20 patients and each patient will be vaccinated with P. vivax-infected red blood cells containing approximately 0.3-1.0 × 10^7 Plasmodium parasites. And successful infection will be indicated by microscopic observation of parasitemia in peripheral blood samples. The treatment will last 3-6 months from the day of successful infection and will be terminated by antimalarial drugs.
  Interventions: Biological: Blood-stage infection of P.vivax

INTERVENTIONS:
Biological: Blood-stage infection of P.vivax — The P. vivax infected blood will be confirmed to follow the national standard of blood donation to ensure that only P. vivax is included, excluding the presence of P. falciparum. Exclude other infectious diseases according to the test of national standard of blood donation.

SUMMARY:
The purpose of this study is to evaluate the safety of Plasmodium immunotherapy and preliminarily evaluate the effectiveness of Plasmodium immunotherapy for advanced cancers.The treatment will last 3-6 months from the day of successful infection and will be terminated by antimalarial drugs.

DETAILED DESCRIPTION:
This study is to enroll 20 patients. Each patient will be vaccinated with P. vivax-infected red blood cells containing approximately 0.3-1.0 × 10^7 Plasmodium parasites and be observed for the exact infection time, parasitemia condition and infection course; principal clinical symptoms such as fever; gastrointestinal reaction; peripheral blood parameters;heart, liver and kidney function; changes in lung function, and dynamic changes in the function of peripheral immune cells. Moreover, the tolerance of patients to Plasmodium infection and changes in tumor-related parameters will be observed preliminarily.The duration of the planned treatment of each subject is 3-6 months. Since the successful infection will be indicated by microscopic observation of parasitemia in peripheral blood samples, the time of the treatment course is based on the presence of peripheral parasitemia. After 3-6 months, parasitemia will be terminated by antimalarial drugs for terminating the treatment of Plasmodium immunotherapy ( the immunological treatment effect may persist after the termination of Plasmodium infection).

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years of age, male or female.
* Patients with advanced cancer confirmed by histopathology and imaging; and imaging lesions of the tumor are clear and measurable, including but not limited to colon cancer, breast cancer, liver cancer, lung cancer, gastric cancer,sarcoma and other solid tumors (except for nasopharyngeal carcinoma, lymphatic cancer, cervical cancer and melanoma).
* The time interval of the termination of chemotherapy (including interventional chemotherapy) or radiotherapy is at least 3 months for patients who had received chemotherapy (including interventional chemotherapy) or radiotherapy; at least 5 half-life for patients who had received targeted drug therapy (the half-life of targeted drug is according to the drug instructions);
* All the patients who have not received surgery, radiotherapy, chemotherapy or targeted drug therapy and refuse to accept the above treatments must meet all the remaining requirements that listed in the inclusion criteria;
* ECGO score of 0 or 1;
* Expected survival ≥ 6 months;
* PLT ≥100× 10^9/L, NE ≥ 1.5 × 10^9/L, and HGB ≥ 100 g/L; no significant morphological abnormalities of red blood cells, or anemia (iron deficiency anemia, autoimmune hemolytic anemia, thalassemia, etc.);
* The peripheral blood count of immune cells is close to normal or normal, the immune function test result is close to or at the level of normal population, and the function of heart, lung, liver and kidney are basically normal (the liver function classification of Child-push is A or B, Cr≤1.5×ULN);
* Patient compliance meets the need for follow-up;
* The subjects are able to understand and sign informed consent.

Exclusion Criteria:

* Patients with severe hemoglobin disease or severe G6PD deficiency;
* Patients with splenectomy or splenomegaly;
* Patients with drug addiction or alcohol dependence;
* With the following diseases or conditions: newly diagnosed with CNS metastasis ( excluding that the tumor lesions of the CNS has disappeared after treatment) and serious or uncontrolled systemic disease or any unstable systemic diseases (including but not limited to active infection, grade three hypertension, unstable angina, congestive heart failure, class III or IV heart disease, severe arrhythmia, liver and kidney dysfunction or metabolic disease), a clear history of neurological or psychiatric disorders, etc;
* Accept any other anti-tumor treatment at the same time;
* Patients with significantly lower immune function than those in the normal population;
* Lung function is seriously damaged, the MNW <39% or can't get out of bed, still feel short of breath when resting;
* Rough cough, dyspnea, without normal diet or difficult to cooperate;
* Poor body condition, the researchers assess that the patients can't tolerate the immune therapy;
* Pregnant or lactating women;
* Women of childbearing age with positive result for pregnancy tests;
* Any condition that makes the subject ineligible to participate (in the opinion of the investigator).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-11-23 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by NCI CTCAE 4.0 | 2 years
  Adverse events will be evaluated according to NCI CTCAE 4.0, and the incidence of adverse events will be calculated.

SECONDARY OUTCOMES:
Progression free survival | 2 years
  Progression free survival (PFS): Starting from treatment until the disease progression is first found or the time of any cause of death (disease progression refers to tumor growth, or metastasis of primary tumor, or discovery of new lesions).
Overall survival | 2 years
  The time starting from the treatment to death of whatever causes (when subjects have lost for follow-up before death, the last follow-up time will be calculated as the time of death).
Tumor marker level | 2 years
  The patient's sensitive tumor markers will be reviewed periodically from the time they are enrolled into the study.
Objective response rate (ORR) | 2 years
  The proportion of patients whose tumor is reduced to a certain amount and maintain a certain period of time.
the Score of Quality of life | 2 years
  Patients are regularly filled with QLQ-C30 (cancer patient quality of life scale) to assess the quality of life of the patients.
1 year of survival rate | 2 years
  The number of cancer cases remaining after 1 year of treatment / the total number of cancer cases treated * 100%.
2 year of survival rate | 2 years
  The number of cancer cases remaining after 2 years of treatment / the total number of cancer cases treated * 100%.
Immunological index | 2 years
  Detection of absolute number of immune cells（such as CD3+CD4+、CD3+CD8+ and so on ）in peripheral blood by flow cytometry.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Fuda Tumor Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Chen L, He Z, Qin L, Li Q, Shi X, Zhao S, Chen L, Zhong N, Chen X. Antitumor effect of malaria parasite infection in a murine Lewis lung cancer model through induction of innate and adaptive immunity. PLoS One. 2011;6(9):e24407. doi: 10.1371/journal.pone.0024407. Epub 2011 Sep 9. PMID 21931708
- [Result] Qin L, Chen C, Chen L, Xue R, Ou-Yang M, Zhou C, Zhao S, He Z, Xia Y, He J, Liu P, Zhong N, Chen X. Worldwide malaria incidence and cancer mortality are inversely associated. Infect Agent Cancer. 2017 Feb 14;12:14. doi: 10.1186/s13027-017-0117-x. eCollection 2017. PMID 28228842
- [Result] Yang Y, Liu Q, Lu J, Adah D, Yu S, Zhao S, Yao Y, Qin L, Qin L, Chen X. Exosomes from Plasmodium-infected hosts inhibit tumor angiogenesis in a murine Lewis lung cancer model. Oncogenesis. 2017 Jun 26;6(6):e351. doi: 10.1038/oncsis.2017.52. PMID 28650446
- [Result] Liu Q, Yang Y, Tan X, Tao Z, Adah D, Yu S, Lu J, Zhao S, Qin L, Qin L, Chen X. Plasmodium parasite as an effective hepatocellular carcinoma antigen glypican-3 delivery vector. Oncotarget. 2017 Apr 11;8(15):24785-24796. doi: 10.18632/oncotarget.15806. PMID 28445973
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/21931708
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5307699/
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5519199/
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/28445973